CLINICAL TRIAL: NCT01822561
Title: Eplerenone for Central Serous Chorioretinopathy: A Pilot Study
Brief Title: Eplerenone for Central Serous Chorioretinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEEC-10722
Record Dates: First submitted 2013-03-25; First posted 2013-04-02 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central Serous Chorioretinopathy; Eplerenone; Optical Coherence Tomography; Enhanced Depth Imaging; Subretinal Fluid
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Eplerenone; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eplerenone (Experimental): All patients in this study will receive Eplerenone 50mg once daily for 4 weeks.
  Interventions: Drug: Eplerenone 50mg

INTERVENTIONS:
Drug: Eplerenone 50mg — All patients will receive the same dose of eplerenone.
  Other Names: Inspra (Pfizer); Eplerenone (Generic)

SUMMARY:
* The goal of the study is to examine the short-term effects and safety of a systemic anti-aldosterone medication, eplerenone, in a small group of patients with central serous chorioretinopathy (CSCR).
* There is currently no standard treatment or therapy for either acute or chronic CSCR, a potentially debilitating eye disease.
* There is evidence in both animals and humans that high blood serum corticosteroid levels can cause or worsen CSCR or findings similar to CSCR in the choroid and retina
* Eplerenone, a mineralocorticoid receptor antagonist, has been shown to be of visual and anatomic benefit in a small series of 4 patients with chronic CSCR, suggesting that decreasing mineralocorticoid action in the eye may improve signs and symptoms of CSCR
* The investigators' aim is to evaluate a standardized dose of eplerenone in a controlled prospective fashion for both acute and chronic CSCR.
* The study consists of taking a standard dose of eplerenone, 50mg once daily, for 1 month
* Over the course of the month, patients will be monitored for side effects, as well as visual and anatomical response to the medication

DETAILED DESCRIPTION:
* The investigators hypothesize that aldosterone inhibition with eplerenone will decrease choroidal vessel vasodilation, focal leakage, and choroidal thickness in patients with both acute and chronic CSCR, leading to resolution of subretinal fluid and ultimately an improvement in symptoms.
* Resolution of sub-retinal fluid will be the primary outcome, which can be precisely measured using optical coherence tomography (OCT)
* Secondary outcomes will include: Change in macular thickness measured with OCT, in central macular circle thickness on OCT, change in visual acuity, change in dye leakage characteristics on fluorescein angiography, change in OCT characteristics of the fellow eye, and safety and tolerability characteristics
* In acute CSCR, subretinal fluid often resolves on its own, but it often takes several months (the literature shows that ~20% of patients have complete resolution of sub-retinal fluid on OCT 1 month after presentation)
* Chronic CSCR is defined as persistent fluid on OCT after 3 months of symptom onset, or recurrence of signs and symptoms within 1 year after the prior episode
* In this study, the investigators will not make a distinction between acute and chronic CSCR
* Eplerenone, a generic medication, is a potassium sparing diuretic, which is FDA approved to treat heart failure as well as high blood pressure, but is not FDA approved for treatment of central serous chorioretinopathy.
* The most important side effect of eplerenone is elevation of serum potassium and decrease of blood pressure
* Patients will therefore be screened with routine blood tests as suggested by the package insert of the medication, and serum potassium and blood pressure will be monitored routinely as directed by the medication package insert
* Study visits will be performed at therapy initiation, 1 week, 2 weeks, and 4 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or over
2. Ability to give written informed consent
3. Presence of sub-retinal fluid under the fovea as seen on OCT
4. Diagnosis of Acute or Chronic CSCR:

   * Acute CSCR: First presentation to eye clinic with visual symptoms, including decreased vision or visual distortion, and the characteristic appearance of CSCR on examination, fluorescein angiography, and OCT.
   * Chronic CSCR: Previous diagnosis of CSCR, persistent subretinal fluid on OCT for more than 3 months after initial presentation to the eye clinic, and <50% reduction in fluid thickness on OCT after 3 months. Patients who have had previous treatment for CSCR may be included.

Exclusion Criteria:

1. Age less than 18
2. Persons with impaired decision-making ability.
3. Women who are known to be pregnant or are actively trying to conceive.
4. Additional eye disease affecting the macula or posterior retina.
5. At screening, serum potassium concentration ≥5.0 mEq/L , a serum creatinine concentration >2 mg/dL in men and >1.8 mg/dL in women, or a creatinine clearance <50 mL/min, and during concomitant administration of potassium supplements, potassium-sparing diuretics, and/or potent CYP3A4 inhibitors (amifostine, cyclosporine, fluconazole, itraconazole, ketoconazole, mifepristone, posaconazole, potassium salts, Rituximab, tacrolimus or voriconazole).
6. Patients with type 2 diabetes will be screened for microalbuminuria with a urinalysis. If microalbuminuria is present, these patients will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre J Witkin, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- New England Eye Center / Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhao M, Celerier I, Bousquet E, Jeanny JC, Jonet L, Savoldelli M, Offret O, Curan A, Farman N, Jaisser F, Behar-Cohen F. Mineralocorticoid receptor is involved in rat and human ocular chorioretinopathy. J Clin Invest. 2012 Jul;122(7):2672-9. doi: 10.1172/JCI61427. Epub 2012 Jun 11. PMID 22684104
- [Background] Gemenetzi M, De Salvo G, Lotery AJ. Central serous chorioretinopathy: an update on pathogenesis and treatment. Eye (Lond). 2010 Dec;24(12):1743-56. doi: 10.1038/eye.2010.130. Epub 2010 Oct 8. PMID 20930852
- [Background] Bouzas EA, Karadimas P, Pournaras CJ. Central serous chorioretinopathy and glucocorticoids. Surv Ophthalmol. 2002 Sep-Oct;47(5):431-48. doi: 10.1016/s0039-6257(02)00338-7. PMID 12431693
- [Background] Chan WM, Lai TY, Lai RY, Liu DT, Lam DS. Half-dose verteporfin photodynamic therapy for acute central serous chorioretinopathy: one-year results of a randomized controlled trial. Ophthalmology. 2008 Oct;115(10):1756-65. doi: 10.1016/j.ophtha.2008.04.014. Epub 2008 Jun 5. PMID 18538401
- [Background] Imamura Y, Fujiwara T, Margolis R, Spaide RF. Enhanced depth imaging optical coherence tomography of the choroid in central serous chorioretinopathy. Retina. 2009 Nov-Dec;29(10):1469-73. doi: 10.1097/IAE.0b013e3181be0a83. PMID 19898183
- [Background] Reibaldi M, Cardascia N, Longo A, Furino C, Avitabile T, Faro S, Sanfilippo M, Russo A, Uva MG, Munno F, Cannemi V, Zagari M, Boscia F. Standard-fluence versus low-fluence photodynamic therapy in chronic central serous chorioretinopathy: a nonrandomized clinical trial. Am J Ophthalmol. 2010 Feb;149(2):307-315.e2. doi: 10.1016/j.ajo.2009.08.026. Epub 2009 Nov 6. PMID 19896635
- [Background] Robertson DM, Ilstrup D. Direct, indirect, and sham laser photocoagulation in the management of central serous chorioretinopathy. Am J Ophthalmol. 1983 Apr;95(4):457-66. doi: 10.1016/0002-9394(83)90265-9. PMID 6682293
- [Background] Nielsen JS, Jampol LM. Oral mifepristone for chronic central serous chorioretinopathy. Retina. 2011 Oct;31(9):1928-36. doi: 10.1097/IAE.0b013e31821c3ef6. PMID 21878843
- [Background] Forooghian F, Meleth AD, Cukras C, Chew EY, Wong WT, Meyerle CB. Finasteride for chronic central serous chorioretinopathy. Retina. 2011 Apr;31(4):766-71. doi: 10.1097/IAE.0b013e3181f04a35. PMID 21273946
- [Background] Weinberger MH, Roniker B, Krause SL, Weiss RJ. Eplerenone, a selective aldosterone blocker, in mild-to-moderate hypertension. Am J Hypertens. 2002 Aug;15(8):709-16. doi: 10.1016/s0895-7061(02)02957-6. PMID 12160194
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Result] Fujimoto H, Gomi F, Wakabayashi T, Sawa M, Tsujikawa M, Tano Y. Morphologic changes in acute central serous chorioretinopathy evaluated by fourier-domain optical coherence tomography. Ophthalmology. 2008 Sep;115(9):1494-500, 1500.e1-2. doi: 10.1016/j.ophtha.2008.01.021. Epub 2008 Apr 18. PMID 18394706
- [Derived] Moein HR, Bierman LW, Novais EA, Moreira-Neto C, Baumal CR, Rogers A, Duker JS, Witkin AJ. Short-term eplerenone for treatment of chronic central serous chorioretinopathy; a prospective study. Int J Retina Vitreous. 2019 Sep 9;5:39. doi: 10.1186/s40942-019-0190-y. eCollection 2019. PMID 31516734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with central serous chorioretinopathy were recruited in the ophthalmology clinic at Tufts Medical Center in Boston, MA between April 2013 and April 2017.
Units Other Than Participants: One eye from each subject was used
Groups:
- Eplerenone Group: All patients in this study received Eplerenone 50mg once daily for 4 weeks.
  Eplerenone 50mg: All patients received the same dose of eplerenone.
Period: Overall Study
Arm/Group | Eplerenone Group
Started | 15; 15 One eye from each subject was used
Completed | 13; 13 One eye from each subject was used
Not Completed | 2; 2 One eye from each subject was used
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 2 Acute CSCR, 11 Chronic CSCR
Groups:
- CSCR Patients Who Received Eplerenone: All patients were diagnosed with central serous chorioretinopathy. All patients received 50mg oral eplerenone daily for 4 weeks.
Arm/Group | CSCR Patients Who Received Eplerenone
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Patients with chronic CSCR [Count of Participants; unit: Participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Complete Resolution of Subretinal Fluid
Description: Optical coherence tomography is an imaging technique capable of extremely high resolution (~5-7 microns) imaging of the macula, and is able to detect the presence and amount of subretinal fluid present, the key anatomic abnormality in Central Serous Chorioretinopathy
Time Frame: Baseline and 1 month after treatment
Measure: Number; unit: participants
Groups:
- Patients That Took Eplerenone: Patients received 50mg oral eplerenone daily for 1 month
Arm/Group | Patients That Took Eplerenone
Number analyzed (Participants) | 13
participants | 0

2. Secondary Outcome: Change in Macular Thickness
Description: Automated software to calculate the thickness of the macula is standard on commercial OCT devices. Macular thickness before and after treatment will be assessed and compared.
Time Frame: Baseline and 1 month after treatment
Measure: Mean (Standard Deviation); unit: Microns
Groups:
- Patients That Received Eplerenone: Patients took 50mg oral eplerenone daily for 1 month
Arm/Group | Patients That Received Eplerenone
Number analyzed (Participants) | 13
Microns | -26 (27)

3. Secondary Outcome: Change in Best Corrected Visual Acuity
Description: Visual acuity will be measured with standard eye charts, with manifest refraction at the initiation and conclusion of treatment. Although an important measure, this was not chosen as the primary outcome measure, as some patients with central serous chorioretinopathy may have a normal visual acuity when properly refracted (refraction can change with elevation of the macula by sub-retinal fluid)
Time Frame: Baseline and 1 month after treatment
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Patients That Took Eplerenone: Patients received oral Eplerenone 50mg once daily for 4 weeks.
Arm/Group | Patients That Took Eplerenone
Number analyzed (Participants) | 13
logMAR | -0.03 (0.08)

4. Secondary Outcome: Change in Subfoveal Choroidal Thickness, Study Eye
Description: Choroidal thickness can be measured using optical coherence tomography, and is known to be affected in patients with central serous chorioretinopathy. Thickness of the choroid under the fovea will be manually calculated in both the study eye.
Time Frame: Baseline and 1 month after treatment
Measure: Mean (Standard Deviation); unit: microns
Groups:
- Patients That Received Eplerenone: Patients received oral Eplerenone 50mg once daily for 4 weeks.
Arm/Group | Patients That Received Eplerenone
Number analyzed (Participants) | 13
microns | 29.8 (18.5)

5. Secondary Outcome: Change in Serum Potassium
Description: Eplerenone can cause elevation of serum potassium. After initial screening, serum potassium was evaluated at 1 and 4 weeks after baseline.
Time Frame: Baseline and 1 month after treatment
Measure: Mean (Standard Deviation); unit: mEq/L
Groups:
- Patients That Received Eplerenone: Patients took oral Eplerenone 50mg once daily for 4 weeks.
Arm/Group | Patients That Received Eplerenone
Number analyzed (Participants) | 13
mEq/L | 0.11 (0.09)

ADVERSE EVENTS:
Time Frame: 3 months. Patients were followed for a minimum of 3 months after treatment was initiated.
Groups:
- Eplerenone Group: All patients had central serous chorioretinopathy and were treated with 50mg oral eplerenone once daily
Arm/Group | Eplerenone Group
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eplerenone Group (N=15)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — One patient stopped treatment after 2 weeks because of subjective shortness of breath. Symptoms resolved within 1 day of stopping the medication.
Palpitations (Cardiac disorders) | 1 (1) — One patient stopped treatment after experiencing subjective headache and heart palpitations after a single dose. Symptoms resolved within 1 day of stopping the medication.

LIMITATIONS AND CAVEATS:
The study had limited enrollment due to lack of interest on the part of potential study subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT01822561/Prot_SAP_000.pdf